CLINICAL TRIAL: NCT00760955
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging, Study to Evaluate the Efficacy and Safety of 3 Doses of TAK-583 in Subjects With Mild to Moderate Diabetic Peripheral Neuropathy
Brief Title: Efficacy and Safety of TAK-583 in Subjects With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-583-006; U1111-1129-7781 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Neuropathies
Keywords: Asymmetric Diabetic Proximal Motor Neuropathy; Diabetic Amyotrophy; Diabetic Autonomic Neuropathy; Diabetic Polyneuropathy; Neuralgia, Diabetic; Symmetric Diabetic Proximal Motor Neuropathy; Drug Therapy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TAK-583 5 mg QD (Experimental)
  Interventions: Drug: TAK-583
- TAK-583 50 mg QD (Experimental)
  Interventions: Drug: TAK-583
- TAK-583 100 mg QD (Experimental)
  Interventions: Drug: TAK-583
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-583 — TAK-583 5 mg, tablets, orally, once daily for up to 6 months.
  Arms: TAK-583 5 mg QD
Drug: TAK-583 — TAK-583 50 mg, tablets, orally, once daily for up to 6 months.
  Arms: TAK-583 50 mg QD
Drug: TAK-583 — TAK-583 100 mg, tablets, orally, once daily for up to 6 months.
  Arms: TAK-583 100 mg QD
Drug: Placebo — TAK-583 placebo-matching tablets, orally, once daily for up to 6 months.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of TAK-583, once daily (QD), in the treatment of neuropathy caused by diabetes mellitus.

DETAILED DESCRIPTION:
Diabetic polyneuropathy is a frequent complication in individuals with type 1 and 2 diabetes mellitus, and can result in progressive functional and structural deficits in both somatic and autonomic nerves. Diabetic polyneuropathy is characterized by degenerative changes in nerve fibers resulting in progressive functional and structural deficits in both somatic and autonomic nerves.

TAK-583 is a synthetic compound currently under development for the treatment of diabetic polyneuropathy. The purpose of this study is to evaluate the safety and efficacy of TAK-583 for the treatment of mild to moderate diabetic polyneuropathy in subjects with type 1 or type 2 diabetes mellitus. Study participation is anticipated to be about 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be post-menopausal or status post documented hysterectomy and bilateral oophorectomy.
* Has fasting clinical laboratory evaluations within the normal reference range for the testing laboratory, or if not, the results must be deemed not clinically significant by the investigator prior to randomization.
* Has Type 1 or type 2 diabetes, as defined by World Health Organization Criteria.
* Has mild to Moderate Diabetic Peripheral Neuropathy defined as:

  * Confirmed abnormality of at least two nerve conduction velocity parameters as defined by the Neurological Core Laboratory.
  * Sural sensory nerve potential amplitude greater than or equal to 1 μV (microvolt).
* Has glycosylated hemoglobin less than or equal to 10%.
* Is on stable pain medications for at least 3 weeks prior to randomization, if applicable.
* Has a glomerular filtration rate calculated by Modification of Diet in Renal Disease of greater than or equal to 45 mL/min/ body surface area.
* Spot albumin/creatinine ratio of less than 300 mg/g creatinine or 33.9 mg/mmol creatinine.
* Has acceptable clinical laboratory test results as defined by:

  * Hemoglobin Greater than or equal to 9.0 g/dL or 5.58 mmol/L
  * Thyroid stimulating hormone Within normal limits
  * Free T4 index Within normal limits
  * B12 level Within normal limits
* Is willing to follow an American Diabetes Association or similar recommended dietary regimen.

Exclusion Criteria

* Individuals with a history of other neuropathies due to causes other than diabetes such as alcohol abuse, liver or renal disease, uremia, toxic exposure, genetic factors, autoimmune disorders, inflammatory demyelinating diseases, monoclonal gammopathies; or endocrine, metabolic or nutritional disorders.
* Has clinical or electrophysiologic evidence of bilateral carpal tunnel syndrome.
* Has a significant skin abnormality or ulcerative changes in their lower extremities that may interfere with the performance of the study related procedures.
* Has a body mass index greater than 45 kg/m2.
* Participants with uncontrolled hypertension or a systolic blood pressure greater than 160 mm Hg or a diastolic blood pressure of greater than 95 mm Hg.
* Has a history of myocardial infarction, coronary angioplasty or bypass graft, unstable angina pectoris, transient ischemic attacks, clinically significant abnormal electrocardiograms, New York Heart Association Functional Classification III or IV, or documented cerebrovascular accident.
* Has a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval greater than 450 milliseconds).
* Has a history of additional risk factors for Torsades de pointes.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Medications that prolong the QT/QTc interval.
  * Lipoic acid.
  * Linolenic acid (primrose oil).
  * Inositol.
  * Topiramate.
  * Acetyl-L-Carnitine.
  * Nerve growth factors.
  * Capsaicin.
  * CYP3A4 inhibitors (amiodarone, diltiazem, Verapamil)
  * HIV protease inhibitors
  * Itraconazole
  * Ketoconazole
  * macrolide antibiotics
  * CYP 3A4 inducers
* Has an alanine aminotransferase level of greater than 1.5 times upper limit of normal, active liver disease or jaundice or Total bilirubin greater than 1.2 times upper limit of normal.
* Has a 12-hour urinary cortisol test greater than 264 nmol/night (95.6 mcg/night) at screening.
* Has clinically significant (as determined by the investigator) or unstable: pulmonary, gastrointestinal, hepatic, hematologic, musculoskeletal, osteoporosis, osteopenia, or endocrine (other than diabetes mellitus or stably treated hypothyroidism) diseases.
* Has a previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug.
* Has any other serious disease or condition at screening or at randomization that might affect life expectancy or make it difficult to successfully manage and follow the subjects according to the protocol.
* Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Has a known hypersensitivity to a compound related to TAK-583.
* Is currently participating in another investigational study or has participated in an investigational study within the past 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline for a composite measure of Maximal Nerve Conduction Velocity of the Peroneal and Median Motor Nerves and the Median and Sural Sensory Nerves. | Month 6 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Electrophysiological Parameters for Individual Nerves. | Month 6 or Final Visit
Change from Baseline in Sensory Sub-Composite and Motor Sub-Composite Scores. | Months 3 and 6 or Final Visit
Change in Vibration Perception Threshold. | Months 3 and 6 or Final Visit
Change in Pain Scores. | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change in Neurological Examination Score. | Months 3 and 6 or Final Visit
Change in Quality of Life Index Score. | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change in glycosylated hemoglobin. | Months 3 and 6 or Final Visit
Change in fasting plasma glucose. | Months 3 and 6 or Final Visit
Change in fasting insulin. | Months 3 and 6 or Final Visit
Change in Fasting C-peptide. | Months 3 and 6 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (38):
- United States (33):
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Huntington Beach, California
  - La Jolla, California
  - Los Angeles, California
  - Pasadena, California
  - Tustin, California
  - Largo, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Palm Beach Gardens, Florida
  - Sunrise, Florida
  - West Palm Beach, Florida
  - Decatur, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Las Vegas, Nevada
  - Englewood, New Jersey
  - Buffalo, New York
  - Staten Island, New York
  - Greenville, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Canada (5):
  - Vancouver, British Columbia
  - Kingston, Ontario
  - North Bay, Ontario
  - Laval, Quebec
  - Québec, Quebec